CLINICAL TRIAL: NCT03039400
Title: Physiotherapist-guided Home Exercise in Moderate to Severe Multiple Sclerosis
Brief Title: Physiotherapist-guided Home Exercise in Moderate to Severe MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Multiple Sclerosis Society of Canada (Other)
Responsible Party: Principal Investigator, Katherine Knox, Associate Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Bio 16-280
Record Dates: First submitted 2016-12-20; First posted 2017-02-01 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based physio group (Experimental): Those in the web-based physio group will have an individual exercise program set up by a treating physiotherapist on webbasedphysio.com after an initial face-to-face assessment. They will be encouraged to undertake their exercise program at least twice per week and diarize their work. Participants will receive a weekly phone call from their treating physiotherapist for the first two weeks. The treating physiotherapist will review the exercise diary of each participant every two weeks, and remotely alter the participant's exercise program as appropriate, by changing exercises, level of difficulty or number of repetitions.
  Interventions: Behavioral: Physiotherapist-guided home exercise with web-based support
- Standard care group (Active Comparator): Those in the standard care group will have their exercise program explained to them at an initial face-to-face assessment with a treating physiotherapist as per usual care. They will receive a written, home-based exercise program. Participants in the usual care group will also be encouraged to undertake their exercise program at least twice per week, and will be asked to keep an exercise diary, in paper format. Participants in the usual care group will also receive a weekly phone call from the physiotherapist for the first two weeks to check on progress.
  Interventions: Behavioral: Physiotherapist-guided home exercise with standard support

INTERVENTIONS:
Behavioral: Physiotherapist-guided home exercise with web-based support — Those in the web-based physio group will access their exercise program online and will be able to leave messages for their physiotherapist on the platform. Physiotherapists will monitor usage and respond to messages every two weeks.
  Arms: Web-based physio group
Behavioral: Physiotherapist-guided home exercise with standard support — Those in the standard care group will receive a written, home-based exercise program. Participants in the usual care group will be asked to keep an exercise diary, in paper format.
  Arms: Standard care group

SUMMARY:
Physical activity is a crucial component to wellness and is associated with multiple health benefits. Persons with MS may find it challenging to participate in regular physical activity or exercise, which is activity done to improve health and/or fitness. This research will test an innovative web-based intervention to help persons with moderate-to-severe disability manage their condition through a maintenance exercise program with specialized physiotherapist guidance and support. The researchers will examine adherence to the web-based physiotherapy program compared to standard physiotherapy care. Forty-five people with MS will be randomly assigned to the web group or standard care group at a rate of 2:1. Participants in the web group will receive supported and individualized web-based physiotherapy. Participants in the standard care group will receive a written exercise program. Regular participation (adherence) in the exercise programs will be evaluated in both groups over six months. The research will also examine participant satisfaction with the programs, safety, MS symptoms, and physical function. A web-based approach may be widely accessible to persons with MS in their own homes and could support long-term participation in physical activity important to wellness.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with MS
* moderate to severe disability (PDDS 2-7)
* able to access the internet in your current living environment

Exclusion Criteria:

* already doing structured exercise more than once per week
* residing >300km from Saskatoon (unless able to travel to Saskatoon for the appointments)
* unable to understand the intent and process of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Adherence to prescribed exercise program | 6 months
  Measured by number of completed exercise sessions on exercise diary

SECONDARY OUTCOMES:
Injury or fall | 6 months
  Participants will be asked to contact their treating physiotherapist in the event of new pain, injury, or fall.
Multiple Sclerosis Impact Scale (MSIS29 v.2) | 6 months
Godin Leisure Time Exercise Questionnaire (GLTEQ) | 6 months
Grip strength measured on hand dynamometer | 6 months
Timed 25-Foot Walk Test | 6 months
Timed Up and Go | 6 months
FIM (R) instrument | 6 months
  The FIM (R) instrument, data set and impairment codes referenced herein are the property of Uniform Data System for Medical Rehabilitation, a division of UB Foundation Activities, Inc.
Hospital Anxiety and Depression Scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Knox, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Department of Physical Medicine & Rehabilitation, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Result] Donkers SJ, Nickel D, Paul L, Wiegers SR, Knox KB. Adherence to Physiotherapy-Guided Web-Based Exercise for Persons with Moderate-to-Severe Multiple Sclerosis: A Randomized Controlled Pilot Study. Int J MS Care. 2020 Sep-Oct;22(5):208-214. doi: 10.7224/1537-2073.2019-048. Epub 2020 Jan 8. PMID 33177956
- [Derived] Knox KB, Nickel D, Donkers SJ, Paul L. Physiotherapist and participant perspectives from a randomized-controlled trial of physiotherapist-supported online vs. paper-based exercise programs for people with moderate to severe multiple sclerosis. Disabil Rehabil. 2023 Apr;45(7):1147-1153. doi: 10.1080/09638288.2022.2055159. Epub 2022 Mar 28. PMID 35341443